CLINICAL TRIAL: NCT00094900
Title: Continuation of a Pilot Open-Label Study of IL 1 Trap in Adult Subjects With Autoinflammatory Diseases: A Therapeutic Approach to Study Pathogenesis
Brief Title: Interleukin-1 Trap to Treat Autoinflammatory Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050014; 05-AR-0014
Record Dates: First submitted 2004-10-28; First posted 2004-10-28 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Inflammation; Familial Mediterranean Fever; Still's Disease, Adult-Onset
Keywords: Muckle Wells Syndrome; NOMID; Adult Stills Disease; Familial Mediterranean; Treatment Trial/Fever; Autoinflammatory Disease
MeSH Terms: conditions — Inflammation; Familial Mediterranean Fever; Still's Disease, Adult-Onset; Cryopyrin-Associated Periodic Syndromes; Fever | interventions — rilonacept

ARMS (1):
- IL-1 Trap (Experimental)
  Interventions: Drug: IL-1 Trap

INTERVENTIONS:
Drug: IL-1 Trap

SUMMARY:
Autoinflammatory diseases are illnesses characterized by episodes of inflammation that, unlike autoimmune disorders, lack the production of high titer autoantibodies or antigen-specific T cells. There is growing genetic and clinical evidence that Interleukin-1 (IL-1) plays a pathogenic role in several of these diseases. This exploratory study aims to examine the utility of the experimental drug candidate, IL 1 Trap (Regeneron Pharmaceuticals, Inc.) in the treatment of adult subjects with the autoinflammatory disorders Neonatal Onset Multisystem Inflammatory Disease (NOMID), Muckle-Wells Syndrome (MWS), and Familial Cold Autoinflammatory Syndrome (FCAS), Familial Mediterranean Fever (FMF), and adult Still's disease. FMF is associated with mutations in pyrin encoding MEFV. NOMID, MWS and FCAS are associated with mutations in cryopyrin-encoding CIAS1.

This pilot study is designed to address: 1) the utility of IL 1 Trap in the treatment of subjects with diseases known to respond to IL-1 blockade (NOMID/MWS/FCAS) as shown by response to treatment with anakinra [Kineret]; 2) the response to IL-1 blockade of subjects with Adult Still's disease and colchicine-resistant FMF once the efficacy of IL-1 Trap has been established in NOMID/MWS/FCAS subjects; and 3) the biochemistry and genetics of autoinflammatory diseases and IL-1 related inflammation.

IL-1 Trap is a recombinant fusion protein with picomolar affinity for IL-1 and a half-life of approximately 7.5 days in humans. This agent is currently in Phase 2 clinical studies for the treatment of rheumatoid arthritis and initial studies have shown activity against clinical and biochemical indicators of inflammation. Compared with anakinra, this agent may exhibit improved dosing convenience, potential for fewer injection site reactions, and improved efficacy due to the extremely high affinity of IL-1Trap for its target.

In this study, biochemical, genetic, and clinical correlates of autoinflammatory disease will initially be measured at baseline following a withdrawal of any TNF or IL-1 inhibitor medications where applicable. Subjects will receive a course of therapy with IL-1 Trap that is predicted to provide an estimated 3-4 weeks of anti-inflammatory activity. Clinical, biochemical, and genetic correlates of inflammation will be measured at appropriate intervals to ascertain response and to further elucidate disease mechanisms. Subjects will be eligible, based on clinical response, to enter a 1- year extension phase with IL-1 Trap. Those subjects who complete the 1-year extension phase, and maintain improved clinical and laboratory parameters compared to baseline values, may continue to receive study medication at their current dose until the study drug is commercially available.

Investigator comment:

This protocol (from the NIH standpoint) is a continuation of the ongoing protocol 05-AR-0014, with a new change in study sponsor, the NIH replacing Regeneron as sponsor. this protocol therefore still contains background and procedural information that refer to patients with FMF and FCAS and or MWS and Still's disease, however only patients with Still's disease will be newly enrolled from this point on, enrollment for the FCAS and or MWS patients has already been completed and it has been decided to not enroll any more FMF patients because the number of subjects is too low to reach reasonable conclusions, in addition it has been difficult to recruit patients that are eligible. The background section and study procedures have largely been left as in the currently IRB approved protocol.

DETAILED DESCRIPTION:
Autoinflammatory diseases are illnesses characterized by episodes of inflammation that, unlike autoimmune disorders, lack the production of high titer autoantibodies or antigen-specific T cells. There is growing genetic and clinical evidence that Interleukin-1 (IL-1) plays a pathogenic role in several of these diseases. This exploratory study aims to examine the utility of the experimental drug candidate, IL 1 Trap (Regeneron Pharmaceuticals, Inc.) in the treatment of adult subjects with the autoinflammatory disorders Neonatal Onset Multisystem Inflammatory Disease (NOMID), Muckle-Wells Syndrome (MWS), and Familial Cold Autoinflammatory Syndrome (FCAS), Familial Mediterranean Fever (FMF), and adult Still's disease. FMF is associated with mutations in MEFV encoding Pyrin. NOMID, MWS and FCAS are associated with mutations in CIAS1-encoding cryopyrin.

This pilot study is designed to address: 1) the utility of IL 1 Trap in the treatment of subjects with diseases known to respond to IL-1 blockade (NOMID/MWS/FCAS) as shown by response to treatment with anakinra [Kineret]; 2) the response to IL-1 blockade of subjects with Adult Still's disease and colchicine-resistant FMF once the efficacy of IL-1 Trap has been established in NOMID/MWS/FCAS subjects; and 3) the biochemistry and genetics of autoinflammatory diseases and IL-1 related inflammation.

IL-1 Trap is a recombinant fusion protein with picomolar affinity for IL-1 and a half-life of approximately 7.5 days in humans. Our result of the FCAS/MWS part of this study and a multi center phase III study in patients with FCAS/MWS provided the basis for the FDA approval of IL-Trap for the treatment of patients with the CAPS.

In this study, biochemical, genetic, and clinical correlates of autoinflammatory disease will initially be measured at baseline following a withdrawal of any TNF or IL-1 inhibitor medications where applicable. Subjects will receive a course of therapy with IL-1 Trap that is predicted to provide an estimated 3-4 weeks of anti-inflammatory activity. Clinical, biochemical, and genetic correlates of inflammation will be measured at appropriate intervals to ascertain response and to further elucidate disease mechanisms. Subjects will be eligible, based on clinical response, to enter a 1- year extension phase with IL-1 Trap. Those subjects who complete the 1-year extension phase, and maintain improved clinical and laboratory parameters compared to baseline values, may continue to receive study medication at their current dose.

Investigator comment:

This protocol (from the NIH standpoint) is a continuation of the ongoing protocol 05-AR-0014, with a new change in study sponsor, the NIH replacing Regeneron as sponsor. This protocol therefore still contains background and procedural information that refer to patients with FMF and FCAS/MWS and Still's disease, however only patients with Still's disease will be newly enrolled from this point on, enrollment for the FCAS/MWS patients has already been completed and it has been decided to not enroll any more FMF patients because the number of subjects is too low to reach reasonable conclusions, in addition it has been difficult to recruit patients that are eligible. Those Adults Still's patients, who complete the extension phase, and maintain improved clinical and laboratory parameters compared to baseline values, may continue to receive study medication at their current dose. These individuals will have their medication supplied by the manufacturing company, Regeneron, until June 2010. At that time the subjects' health insurance companies will begin to pay for their medication supply or the subjects will begin treatment with Anakinra, another IL-1 blocker. Our follow-up plans for all patients who discontinue IL-1 Trap usage will be to monitor for any medication side effects or toxicities and collect adverse event data for 3 months post discontinuation. We will help our subjects to obtain insurance coverage for IL-1Trap.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male or female subjects with inflammatory disease greater than or equal to 18 years of age.

Participation in NIH study number 94-AR-0105 ("Genetics and Pathophysiology of FMF and Related Disorders")

Subjects presenting with active NOMID, MWS, FCAS, FMF, or adult Still's disease based on clinical signs/symptoms and/or biochemical markers such as acute phase reactants (CRP, SAA or ESR). Subjects need not have both clinical features and biochemical markers of disease to be enrolled. However, both clinical and laboratory responses will be evaluated in each subject for improvement as outcome measures (even improvement of laboratory values found to be within the normal range at baseline).

* NOMID, MWS, and FCAS: Diagnosis will be based on the history of classical features of disease including fevers, rash, joint involvement, CNS involvement. Approximately half of all subjects with these clinical syndromes are mutation negative; however, in the experience of the principal investigator these subjects show favorable clinical response to IL-1 blockade with anakinra. Therefore, subjects with or without recognized mutations in CIAS1 will be eligible to enroll in this study. Active disease will be defined as either the presence of aforementioned classical features, or a history of such features that became quiescent in the setting of therapy with anakinra. However, before a patient who has quiescent disease and is currently taking anakinra can receive study drug, he/she must fulfill criteria for active disease after anakinra has been discontinued.
* FMF will be diagnosed on the basis of documented presence of one or two mutant alleles of MEFV as well as the history of classical clinical features of FMF such as periodic fevers, rash, arthritis, arthralgia, or episodes of serositis. Subjects must be considered non-responsive to colchicine (up to 2 milligrams per day) on the basis of continued symptoms or flares (greater than or equal to one per month) or elevated acute phase reactants (ESR, CRP or SAA greater than or equal to 1.5 times the upper limit of normal between attacks) despite treatment with maximally tolerated doses of colchicine. Positive genetic test will be required for FMF to rule out the possibility that non-response to colchicine is due to misdiagnosis.
* Adult Still's disease will be diagnosed on the basis of history of classical clinical features such as fevers, evanescent salmon-pink rash, arthritis, arthralgia, and myalgia. Active disease will be defined as presence of one or more of these features and/ or elevation of acute phase reactants (ESR, CRP or SAA greater than or equal to 1.5 times the upper limit of normal).
* Subjects currently treated with anakinra may be enrolled in this study even though autoinflammatory disease may be quiescent. For these subjects a history of active autoinflammatory disease prior to treatment with anakinra will be sufficient. Subjects must be greater than 48 hours from their last dose of anakinra before beginning IL-1 Trap therapy, and will not take anakinra for the remainder of their enrollment in the study. However, before study drug is administered subjects have to manifest signs of active disease as described above

Stable dose of steroids, NSAIDs, DMARDs, or colchicine for four weeks prior to enrollment visit.

Females of childbearing potential (young women who have had at least one menstrual period regardless of age) must have a negative urine pregnancy test at screening and a negative serum pregnancy test at baseline prior to performance of any radiologic procedure or administration of study medication.

Women of childbearing age and men able to father a child, who are sexually active, who agree to use a form of effective birth control, including abstinence.

Negative PPD test using 5 T.U. intradermal testing per CDC guidelines, and no evidence of active TB on chest X-ray. Subjects with latent TB (positive PPD test) currently treated with adequate therapy initiated for at least one month prior to first dose of study medication may be included. Full prophylaxis regimens will be completed. Subjects who have been BCG-vaccinated will also be skin-tested.

Able to understand, and complete study-related questionnaires.

Able and willing to give informed consent and abide with the study procedures.

EXCLUSION CRITERIA:

Treatment with a live virus vaccine during 3 months prior to baseline visit. No live vaccines will be allowed throughout the course of this study.

Current treatment with TNF inhibitors or recent discontinuation of TNF inhibitors (use within less than 5 half-lives of TNF inhibitor agent).

Presence of active infections or a history of pulmonary TB infection with or without documented adequate therapy. Subjects with current active TB, or recent close exposure to an individual with active TB are excluded from the study.

Chest x-ray read by a radiologist with pleural scarring and/or calcified granuloma consistent with prior TB.

Positive test for or prior history of HIV, Hepatitis B or C.

History or concomitant diagnosis of congestive heart failure.

History of malignancy. Subjects deemed cured of superficial malignancies such as cutaneous basal or squamous cell carcinomas, or in situ cervical cancer may be enrolled.

Known hypersensitivity to CHO cell derived biologicals or any components of IL 1 Trap.

Presence of any additional rheumatic disease or significant systemic disease. For example, major chronic infectious/ inflammatory/ immunologic disease (such as inflammatory bowel disease, psoriatic arthritis, spondyloarthropathy, SLE in addition to autoinflammatory disease).

Presence of any of the following laboratory abnormalities at enrollment visit: creatinine greater than 1.5 times the upper limit of normal, WBC less than 3.6 x 10(9)/mm(3); platelet count less than 150,000 mm(3); ALT or AST greater than 2.0 x ULN (ALT/AST greater than 2.0 x ULN in an adult Still's disease patient would prompt a hepatology consult prior to enrollment unless these abnormalities are considered by the Principal Investigator to be reflective of the underlying Still's disease).

Lactating females or pregnant females.

Subjects with asthma not adequately controlled on current therapy.

Enrollment in any other investigational treatment study or use of an investigational agent, or has not yet completed at least 4 weeks or 5 half-lives, whichever is longer, since ending another investigational device or drug trial.

Subjects for whom there is concern about compliance with the protocol procedures.

Presence of other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the subject's safety, inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-10; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aksentijevich I, Nowak M, Mallah M, Chae JJ, Watford WT, Hofmann SR, Stein L, Russo R, Goldsmith D, Dent P, Rosenberg HF, Austin F, Remmers EF, Balow JE Jr, Rosenzweig S, Komarow H, Shoham NG, Wood G, Jones J, Mangra N, Carrero H, Adams BS, Moore TL, Schikler K, Hoffman H, Lovell DJ, Lipnick R, Barron K, O'Shea JJ, Kastner DL, Goldbach-Mansky R. De novo CIAS1 mutations, cytokine activation, and evidence for genetic heterogeneity in patients with neonatal-onset multisystem inflammatory disease (NOMID): a new member of the expanding family of pyrin-associated autoinflammatory diseases. Arthritis Rheum. 2002 Dec;46(12):3340-8. doi: 10.1002/art.10688. PMID 12483741
- [Background] Chae JJ, Komarow HD, Cheng J, Wood G, Raben N, Liu PP, Kastner DL. Targeted disruption of pyrin, the FMF protein, causes heightened sensitivity to endotoxin and a defect in macrophage apoptosis. Mol Cell. 2003 Mar;11(3):591-604. doi: 10.1016/s1097-2765(03)00056-x. PMID 12667444
- [Background] De Benedetti F, Pignatti P, Massa M, Sartirana P, Ravelli A, Martini A. Circulating levels of interleukin 1 beta and of interleukin 1 receptor antagonist in systemic juvenile chronic arthritis. Clin Exp Rheumatol. 1995 Nov-Dec;13(6):779-84. PMID 8835254
- [Derived] Goldbach-Mansky R, Shroff SD, Wilson M, Snyder C, Plehn S, Barham B, Pham TH, Pucino F, Wesley RA, Papadopoulos JH, Weinstein SP, Mellis SJ, Kastner DL. A pilot study to evaluate the safety and efficacy of the long-acting interleukin-1 inhibitor rilonacept (interleukin-1 Trap) in patients with familial cold autoinflammatory syndrome. Arthritis Rheum. 2008 Aug;58(8):2432-42. doi: 10.1002/art.23620. PMID 18668591
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-AR-0014.html

RESULTS

PARTICIPANT FLOW:
Groups:
- IL-1 Trap: Subjects received initial dose of 100mg per day for 3 consecutive days and did not receive any more till a disease flare occured
Period: Overall Study
Arm/Group | IL-1 Trap
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Daily Scores
Description: Daily scores change from baseline to 10 days. The clinical daily diary scores (a composite score that included fever, rash, and arthritis/arthralgia, with each of the 3 symptoms scored from 0 [no symptom] to 4 [worst symptom], with an overall range score of 0-12).
Time Frame: 10 days for 4 patient, 6 days for 1 patient
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -3.09 (1.03)

2. Primary Outcome: Mean Change in ESR
Description: ESR change from baseline to 10 days.The Erythrocyte Sedimentation Rate (ESR) is an acute phase reactant measured to evaluate lab parameters of inflammation
Time Frame: 10 days for 4 patient, 6 days for 1 patient
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: mm/hour
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mm/hour | -32.2 (7.31)

3. Primary Outcome: Mean Change in hsCRP
Description: hsCRP change from baseline to 10 days.The high sensitivity C-reactive protein (hsCRP) is an acute phase reactant measured to evaluate lab parameters of inflammation
Time Frame: 10 days for 4 patient, 6 days for 1 patient
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/dl | -4.22 (0.98)

4. Primary Outcome: Mean Change in SAA
Description: SAA change from baseline to 10 days.The serum Amyloid A (SAA) is an acute phase reactant measured to evaluate lab parameters of inflammation
Time Frame: 10 days for 4 patient, 6 days for 1 patient
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: mg/liter
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/liter | -216.1 (92.14)

5. Primary Outcome: Response to Treatment (ACR20) in Patients With Adult Onset Still's Disease
Description: At the 24 month post-dose visit, an ACR20 responder was defined as someone who achieved at least 20% improvement in the tender and the swollen 28-joint count, and 20% improvement in at least 3 of the following 5 measures: Patient's pain assessment, Patient's global assessment of disease activity, Physician's global assessment of disease activity, Patient self-assessed disability, Acute phase reactant.
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Number; unit: participants
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
participants | 3

6. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS
Description: Patient's global assessment change by visual analog scale from baseline to 3 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 3 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -5.29 (0.67)

7. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS
Description: Patient's global assessment change by visual analog scale from baseline to 6 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 6 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -2.56 (1.27)

8. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS
Description: Patient's global assessment change by visual analog scale from baseline to 9 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 9 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -2.63 (1.19)

9. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS
Description: Patient's global assessment change by visual analog scale from baseline to 12 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 12 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -2.86 (1.24)

10. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS
Description: Patient's global assessment change by visual analog scale from baseline to 16 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 16 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -3.40 (0.98)

11. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS
Description: Patient's global assessment change by visual analog scale from baseline to 20 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 20 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -2.78 (1.13)

12. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS
Description: Patient's global assessment change by visual analog scale from baseline to 24 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 24 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -2.33 (1.3)

13. Secondary Outcome: Mean Change in Physician's Global Assessment, by VAS
Description: Physician's global assessment change by visual analog scale from baseline to 3 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 3 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -4.15 (0.89)

14. Secondary Outcome: Mean Change in Physician's Global Assessment, by VAS
Description: Physician's global assessment change by visual analog scale from baseline to 6 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 6 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -4.27 (1.01)

15. Secondary Outcome: Mean Change in Physician's Global Assessment, by VAS
Description: Physician's global assessment change by visual analog scale from baseline to 9 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 9 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -4.71 (0.75)

16. Secondary Outcome: Mean Change in Physician's Global Assessment, by VAS
Description: Physician's global assessment change by visual analog scale from baseline to 12 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 12 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -4.30 (0.9)

17. Secondary Outcome: Mean Change in Physician's Global Assessment, by VAS
Description: Physician's global assessment change by visual analog scale from baseline to 16 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 16 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -4.85 (0.95)

18. Secondary Outcome: Mean Change in Physician's Global Assessment, by VAS
Description: Physician's global assessment change by visual analog scale from baseline to 20 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 20 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -4.79 (0.66)

19. Secondary Outcome: Mean Change in Physician's Global Assessment, by VAS
Description: Physician's global assessment change by visual analog scale from baseline to 24 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 24 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -4.54 (0.99)

20. Secondary Outcome: Mean Change in Patient's Assessment of Pain, by VAS
Description: Patient's global assessment of pain by visual analog scale from baseline to 3 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 3 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -5.43 (1.2)

21. Secondary Outcome: Mean Change in Patient's Assessment of Pain, by VAS
Description: Patient's global assessment of pain by visual analog scale from baseline to 6 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 6 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -4.24 (1.24)

22. Secondary Outcome: Mean Change in Patient's Assessment of Pain, by VAS
Description: Patient's global assessment of pain by visual analog scale from baseline to 9 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 9 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -3.93 (1.28)

23. Secondary Outcome: Mean Change in Patient's Assessment of Pain, by VAS
Description: Patient's global assessment of pain by visual analog scale from baseline to 12 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 12 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -3.08 (2.28)

24. Secondary Outcome: Mean Change in Patient's Assessment of Pain, by VAS
Description: Patient's global assessment of pain by visual analog scale from baseline to 16 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 16 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -5.65 (1.13)

25. Secondary Outcome: Mean Change in Patient's Assessment of Pain, by VAS
Description: Patient's global assessment of pain by visual analog scale from baseline to 20 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 20 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -5.01 (1.22)

26. Secondary Outcome: Mean Change in Patient's Assessment of Pain, by VAS
Description: Patient's global assessment of pain by visual analog scale from baseline to 24 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 24 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -4.82 (1.22)

27. Secondary Outcome: Mean Change in Patient's Assessment of Fatigue, by VAS
Description: Patient's assessment of fatigue by visual analog scale from baseline to 3 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 3 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -3.12 (1.04)

28. Secondary Outcome: Mean Change in Patient's Assessment of Fatigue, by VAS
Description: Patient's assessment of fatigue by visual analog scale from baseline to 6 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 6 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -2.27 (1.15)

29. Secondary Outcome: Mean Change in Patient's Assessment of Fatigue, by VAS
Description: Patient's assessment of fatigue by visual analog scale from baseline to 9 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 9 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -2.41 (1.1)

30. Secondary Outcome: Mean Change in Patient's Assessment of Fatigue, by VAS
Description: Patient's assessment of fatigue by visual analog scale from baseline to 12 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 12 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -2.04 (1.17)

31. Secondary Outcome: Mean Change in Patient's Assessment of Fatigue, by VAS
Description: Patient's assessment of fatigue by visual analog scale from baseline to 16 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 16 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -3.16 (0.67)

32. Secondary Outcome: Mean Change in Patient's Assessment of Fatigue, by VAS
Description: Patient's assessment of fatigue by visual analog scale from baseline to 20 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 20 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -2.38 (0.89)

33. Secondary Outcome: Mean Change in Patient's Assessment of Fatigue, by VAS
Description: Patient's assessment of fatigue by visual analog scale from baseline to 24 months. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The VAS had a range of 0-10 cm, with 0 as none and 10 being the worst.
Time Frame: 24 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -3.19 (1.63)

34. Secondary Outcome: Mean Change in Tender Joint Count
Description: Count of tender joints in patient from baseline to 3 months. 68 tender joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 3 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -5.70 (3.49)

35. Secondary Outcome: Mean Change in Tender Joint Count.
Description: Count of tender joints in patient from baseline to 6 months. 68 tender joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 6 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -4.30 (4.47)

36. Secondary Outcome: Mean Change in Tender Joint Count
Description: Count of tender joints in patient from baseline to 9 months. 68 tender joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 9 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -4.80 (4.73)

37. Secondary Outcome: Mean Change in Tender Joint Count
Description: Count of tender joints in patient from baseline to 12 months. 68 tender joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 12 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -7.40 (5.33)

38. Secondary Outcome: Mean Change in Tender Joint Count
Description: Count of tender joints in patient from baseline to 16 months. 68 tender joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 16 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -9.60 (5.71)

39. Secondary Outcome: Mean Change in Tender Joint Count
Description: Count of tender joints in patient from baseline to 20 months. 68 tender joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 20 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -8.40 (4.77)

40. Secondary Outcome: Mean Change in Tender Joint Count
Description: Count of tender joints in patient from baseline to 24 months. 68 tender joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 24 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -6.80 (5.53)

41. Secondary Outcome: Mean Change in Swollen Joint Count
Description: Count of swollen joints in patient from baseline to 3 months. 68 swollen joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 3 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | -7.90 (4.64)

42. Secondary Outcome: Mean Change in Swollen Joint Count
Description: Count of swollen joints in patient from baseline to 6 months. 68 swollen joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 6 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | -2.50 (3.66)

43. Secondary Outcome: Mean Change in Swollen Joint Count
Description: Count of swollen joints in patient from baseline to 9 months. 68 swollen joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 9 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | -2.30 (3.33)

44. Secondary Outcome: Mean Change in Swollen Joint Count
Description: Count of swollen joints in patient from baseline to 12 months. 68 swollen joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 12 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | -6.10 (2.82)

45. Secondary Outcome: Mean Change in Swollen Joint Count
Description: Count of swollen joints in patient from baseline to 16 months. 68 swollen joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 16 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | -9.00 (4.09)

46. Secondary Outcome: Mean Change in Swollen Joint Count
Description: Count of swollen joints in patient from baseline to 20 months. 68 swollen joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 20 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | -9.40 (3.59)

47. Secondary Outcome: Mean Change in Swollen Joint Count
Description: Count of swollen joints in patient from baseline to 24 months. 68 swollen joints were assessed manually in a standardized fashion. (Reference: Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995;38:727.-35)
Time Frame: 24 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | -4.20 (4.45)

48. Secondary Outcome: Mean Change in SF-36 Physical Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), physical component score, taken by patient from baseline to 3 months. Lower scores indicate limited physical function, while higher scores indicate higher physical function. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection. Med Care 1992;30:473-83.)
Time Frame: 3 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 11.11 (3.74)

49. Secondary Outcome: Mean Change in SF-36 Physical Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), physical component score, taken by patient from baseline to 6 months. Lower scores indicate limited physical function, while higher scores indicate higher physical function. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection. Med Care 1992;30:473-83.)
Time Frame: 6 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 13.09 (3.19)

50. Secondary Outcome: Mean Change in SF-36 Physical Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), physical component score, taken by patient from baseline to 9 months. Lower scores indicate limited physical function, while higher scores indicate higher physical function. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection. Med Care 1992;30:473-83.)
Time Frame: 9 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 10.38 (4.45)

51. Secondary Outcome: Mean Change in SF-36 Physical Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), physical component score, taken by patient from baseline to 12 months. Lower scores indicate limited physical function, while higher scores indicate higher physical function. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection. Med Care 1992;30:473-83.)
Time Frame: 12 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 13.28 (3.84)

52. Secondary Outcome: Mean Change in SF-36 Physical Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), physical component score, taken by patient from baseline to 16 months. Lower scores indicate limited physical function, while higher scores indicate higher physical function. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection. Med Care 1992;30:473-83.)
Time Frame: 16 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 12.58 (3.23)

53. Secondary Outcome: Mean Change in SF-36 Physical Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), physical component score, taken by patient from baseline to 20 months. Lower scores indicate limited physical function, while higher scores indicate higher physical function. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection. Med Care 1992;30:473-83.)
Time Frame: 20 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 10.12 (5.48)

54. Secondary Outcome: Mean Change in SF-36 Physical Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), physical component score, taken by patient from baseline to 24 months. Lower scores indicate limited physical function, while higher scores indicate higher physical function. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection. Med Care 1992;30:473-83.)
Time Frame: 24 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 10.22 (4.59)

55. Secondary Outcome: Mean Change in SF-36 Mental Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), mental component score, taken by patient from baseline to 3 months. Lower scores indicate feeling depressed, anxious all the time, while higher scores indicate a state of happiness and peacefulness. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection.Med Care 1992;30:473-83.)
Time Frame: 3 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 7.56 (4.97)

56. Secondary Outcome: Mean Change in SF-36 Mental Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), mental component score, taken by patient from baseline to 6 months. Lower scores indicate feeling depressed, anxious all the time, while higher scores indicate a state of happiness and peacefulness. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection.Med Care 1992;30:473-83.)
Time Frame: 6 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 5.95 (4.01)

57. Secondary Outcome: Mean Change in SF-36 Mental Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), mental component score, taken by patient from baseline to 9 months. Lower scores indicate feeling depressed, anxious all the time, while higher scores indicate a state of happiness and peacefulness. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection.Med Care 1992;30:473-83.)
Time Frame: 9 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 8.8 (4)

58. Secondary Outcome: Mean Change in SF-36 Mental Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), mental component score, taken by patient from baseline to 12 months. Lower scores indicate feeling depressed, anxious all the time, while higher scores indicate a state of happiness and peacefulness. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection.Med Care 1992;30:473-83.)
Time Frame: 12 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 9.76 (3.46)

59. Secondary Outcome: Mean Change in SF-36 Mental Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), mental component score, taken by patient from baseline to 16 months. Lower scores indicate feeling depressed, anxious all the time, while higher scores indicate a state of happiness and peacefulness. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection.Med Care 1992;30:473-83.)
Time Frame: 16 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 11.74 (6.42)

60. Secondary Outcome: Mean Change in SF-36 Mental Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), mental component score, taken by patient from baseline to 20 months. Lower scores indicate feeling depressed, anxious all the time, while higher scores indicate a state of happiness and peacefulness. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection.Med Care 1992;30:473-83.)
Time Frame: 20 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 12.98 (3.96)

61. Secondary Outcome: Mean Change in SF-36 Mental Component Score
Description: Short Form 36 health survey (range 0-100 for each component score), mental component score, taken by patient from baseline to 24 months. Lower scores indicate feeling depressed, anxious all the time, while higher scores indicate a state of happiness and peacefulness. (Reference: Ware JE Jr, Sherbourne CD. The MOS 36-item Short-Form health survey (SF-36). I. Conceptual framework and item selection.Med Care 1992;30:473-83.)
Time Frame: 24 months
Population: The analyses included only those subjects with Familial Cold Autoinflammatory Syndrome (FCAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | 11.46 (6.46)

62. Secondary Outcome: Mean Change in WBCs
Description: White Blood Cell count change from baseline to 3 months
Time Frame: 3 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: x 10^3 cells/microliter
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
x 10^3 cells/microliter | 0.57 (1.17)

63. Secondary Outcome: Mean Change in WBCs
Description: White Blood Cell count change from baseline to 6 months
Time Frame: 6 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: x 10^3 cells/microliter
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
x 10^3 cells/microliter | -1.29 (1.35)

64. Secondary Outcome: Mean Change in WBCs
Description: White Blood Cell count change from baseline to 12 months
Time Frame: 12 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: x 10^3 cells/microliter
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
x 10^3 cells/microliter | -0.87 (1.08)

65. Secondary Outcome: Mean Change in WBCs
Description: White Blood Cell count change from baseline to 24 months
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: x 10^3 cells/microliter
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
x 10^3 cells/microliter | -2.88 (1.43)

66. Secondary Outcome: Mean Change in Ferritin
Description: Ferritin level change from baseline to 3 months
Time Frame: 3 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mcg/L | -231.80 (138.11)

67. Secondary Outcome: Mean Change in Ferritin
Description: Ferritin level change from baseline to 6 months
Time Frame: 6 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mcg/L | -184.80 (88.19)

68. Secondary Outcome: Mean Change in Ferritin
Description: Ferritin level change from baseline to 12 months
Time Frame: 12 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mcg/L | 331.80 (575.34)

69. Secondary Outcome: Mean Change in Ferritin
Description: Ferritin level change from baseline to 24 months
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mcg/L | -263.80 (114.69)

70. Secondary Outcome: Mean Change in Serum Amyloid A
Time Frame: 3 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/liter
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/liter | -117.80 (62.54)

71. Secondary Outcome: Mean Change in Serum Amyloid A
Time Frame: 6 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/liter
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/liter | -173.40 (80.56)

72. Secondary Outcome: Mean Change in Serum Amyloid A
Time Frame: 12 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/liter
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/liter | -274.20 (103.18)

73. Secondary Outcome: Mean Change in Serum Amyloid A
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/liter
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/liter | -173.25 (115.86)

74. Secondary Outcome: Mean Change in C-Reactive Protein
Time Frame: 3 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/dl | -4.79 (2.71)

75. Secondary Outcome: Mean Change in C-Reactive Protein
Time Frame: 6 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/dl | -5.67 (2.62)

76. Secondary Outcome: Mean Change in C-Reactive Protein
Time Frame: 12 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/dl | -7.06 (2.38)

77. Secondary Outcome: Mean Change in C-Reactive Protein
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/dl | -4.91 (1.86)

78. Secondary Outcome: Mean Change in Erythrocyte Sedimentation Rate
Time Frame: 3 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mm/hour
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mm/hour | -13.20 (10.85)

79. Secondary Outcome: Mean Change in Erythrocyte Sedimentation Rate
Time Frame: 6 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mm/hour
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mm/hour | -32.40 (11.12)

80. Secondary Outcome: Mean Change in Erythrocyte Sedimentation Rate
Time Frame: 12 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mm/hour
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mm/hour | -34.60 (14.26)

81. Secondary Outcome: Mean Change in Erythrocyte Sedimentation Rate
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mm/hour
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mm/hour | -23.40 (15.02)

82. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS in AOSD Subjects
Description: as for outcome 6
Time Frame: 3 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -0.16 (0.79)

83. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS in AOSD Subjects
Description: as for outcome 7
Time Frame: 6 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -0.75 (0.60)

84. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS in AOSD Subjects
Description: as for outcome 9
Time Frame: 12 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -0.97 (1.34)

85. Secondary Outcome: Mean Change in Patient's Global Assessment, by VAS in AOSD Subjects
Description: as for outcome 12
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
units on a scale | -1.03 (0.96)

86. Secondary Outcome: Mean Change in Tender Joint Count in AOSD Subjects
Description: as for outcome 34
Time Frame: 3 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | 1.60 (2.98)

87. Secondary Outcome: Mean Change in Tender Joint Count in AOSD Subjects
Description: as for outcome 35
Time Frame: 6 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -2.00 (1.48)

88. Secondary Outcome: Mean Change in Tender Joint Count in AOSD Subjects
Description: as for outcome 37
Time Frame: 12 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -3.40 (3.06)

89. Secondary Outcome: Mean Change in Tender Joint Count in AOSD Subjects
Description: as for outcome 40
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
tender joints | -6.80 (3.28)

90. Secondary Outcome: Mean Change in Swollen Joint Count in AOSD Subjects
Description: as for outcome 41
Time Frame: 3 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | 1.20 (3.89)

91. Secondary Outcome: Mean Change in Swollen Joint Count in AOSD Subjects
Description: as for outcome 42
Time Frame: 6 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | 0.60 (2.79)

92. Secondary Outcome: Mean Change in Swollen Joint Count in AOSD Subjects
Description: as for outcome 44
Time Frame: 12 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | -2.40 (2.60)

93. Secondary Outcome: Mean Change in Swollen Joint Count in AOSD Subjects
Description: as for outcome 47
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
swollen joints | -2.60 (1.81)

94. Secondary Outcome: Mean Change in Prednisone Dose
Time Frame: 3 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/day | -0.50 (1.66)

95. Secondary Outcome: Mean Change in Prednisone Dose
Time Frame: 6 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/day | -1.50 (7.81)

96. Secondary Outcome: Mean Change in Prednisone Dose
Time Frame: 12 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/day | -4.10 (6.52)

97. Secondary Outcome: Mean Change in Prednisone Dose
Time Frame: 24 months
Population: The analyses included only those subjects with Adult Onset Still's Disease (AOSD)
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | IL-1 Trap
Number analyzed (Participants) | 5
mg/day | -7.00 (7.20)

ADVERSE EVENTS:
Arm/Group | IL-1 Trap
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IL-1 Trap (N=11)
Blood and lymphatic system disorders - Other (Macrophage Activation Syndrome) (Blood and lymphatic system disorders) | 1
Joint infection-mycobacterium (Infections and infestations) | 1
Skin Infection-mycobacterium (Infections and infestations) | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1
Kidney infection (Renal and urinary disorders) | 1
Renal Calculi (Renal and urinary disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IL-1 Trap (N=11)
Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic disorder- other (Iron Deficiency) (Blood and lymphatic system disorders) | 1
Ear disorder - congestion (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Endocrine disorder - other (Inhomogeneous thyroid) (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Eye disorder - other (Hordeolum) (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Flu like symptoms (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Bronchial infection (Infections and infestations) | 4
Enterocolitis infectious (Infections and infestations) | 1
Eye Infection (Infections and infestations) | 1
Joint infection (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 2
Mucosal infection (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 7
Skin infection (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 2
upper respiratory infection (Infections and infestations) | 6
Urinary Tract Infection (Infections and infestations) | 2
Vaginal Infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood gonadotrophin abnormal (Investigations) | 1
Cholesterol high (Investigations) | 3
High cholesterol (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
weight gain (Investigations) | 3
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and Connective tissue disorder - other (Flexion contracture) (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and Connective tissue disorder - other (Ruptured Baker's cyst) (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and Connective tissue disorder -other (Bursa fluid) (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and Connective tissue disorder -other (Bursitis) (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and Connective tissue disorder -other (Synovial cyst) (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasm, benign, malignant and unspecified (basal cell carcinoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm, benign, malignant and unspecified (cysts and polyps) - Lung nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm, benign, malignant and unspecified (cysts and polyps) - Pilonidal sinus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Memory Impairment (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Libido decreased (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Renal Calculi (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Irregular Menstruation (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorder - other (Increased skin fold) (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorder - other (skin tear) (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Secondary outcome analyses will be stratified based on primary outcome results - responders and non-responders.

1 subject with Familial Mediterranean Fever (FMF) was recruited but outcomes were not collected due to insufficient accrual of FMF cases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes